CLINICAL TRIAL: NCT01424618
Title: A Novel Approach to Endometrial Preparation in Recipients of Donor Cycles
Brief Title: A Novel Approach to Endometrial Preparation in Recipients of Donor Eggs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kelly, Maureen, M.D. (Individual)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Maureen Kelly, M.D., Medical Director, Kelly, Maureen, M.D.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 39604
Record Dates: First submitted 2011-08-25; First posted 2011-08-29 (Estimated); Last update posted 2011-08-29 (Estimated); Status verified 2011-08

CONDITIONS: Implantation, Embryo
Keywords: Donor eggs; Donor oocytes; Pregnancy; Embryo Implantation; Infertility; IVF
MeSH Terms: conditions — Infertility | interventions — Leuprolide; ganirelix

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GnRh agonist (Active Comparator): This arm will use a GnRH agonist to suppress pituitary-ovarian function
  Interventions: Drug: Leuprolide
- GnRH antagonist (Experimental): A GnRH antagonist will be used to suppress pituitary-ovarian function
  Interventions: Drug: Ganirelix

INTERVENTIONS:
Drug: Leuprolide — leuprolide 10 units daily, decreased to 5 units daily once suppression achieved for a total of approximately 4 weeks. Once suppression achieved, estradiol and progesterone administered to mature uterine lining.
  Other Names: Lupron
  Arms: GnRh agonist
Drug: Ganirelix — Ganirelix 250 mcg daily will be used to suppress pituitary-ovarian function and is administered concurrently with estradiol and progesterone for approximately two weeks.
  Other Names: Antagon
  Arms: GnRH antagonist

SUMMARY:
This study compares two different methods to prepare the uterine lining of recipients for implantation in cycles using donor eggs. The study method requires less time than the standard method.

It is hypothesized that both methods would be suitable for use in egg donor cycles.

DETAILED DESCRIPTION:
Currently a combination of medications is used to prepare the uterine lining of recipients for implantation in egg donor cycles. The protocol used most commonly is as follows: Initially the individual's own pituitary-ovarian system is suppressed using a GnRH agonist so there are not conflicting signals sent to the uterus. This is followed by hormonal medication identical to what is secreted by the ovaries to prepare the uterine lining for subsequent embryo transfer in donor egg cycles.This preparation typically takes a minimum of four weeks.

This study will compare a different medication, a GnRh antagonist (which is commonly used in IVF) to suppress an individual's system during the preparation of the uterine lining. This protocol would generally take only two weeks to prepare the uterine lining.

ELIGIBILITY:
Inclusion Criteria:

* recipients awaiting egg donation
* some ovarian function
* normal endometrial cavity

Exclusion Criteria:

* submucosal myoma
* myoma(s) greater than 4 centimeters
* endometrial polyp
* DES exposure
* documented recalcitrant thin endometrium ( <7 mm)
* untreated vulvovaginitis
* active pelvic infection
* endometrial cancer or suspected/known hormonally sensitive cancers
* breast cancer
* thromboembolic disease
* cerebrovascular or coronary heart disease
* diabetes mellitus
* hepatic tumors or active liver disease
* severe hypertension
* headaches with neurologic disease
* cholestatic disease
* heavy smoking over age 35

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-01; Primary Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
endometrial thickness measured by ultrasound | 2-4 weeks
  In office ultrasound to measure thickness of endometrial lining.

SECONDARY OUTCOMES:
endometrial biopsy | 3-6 weeks
  In office aspiration of endometrial cells will be examined microscopically to determine if they are at an appropriate stage for implantation.

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Kelly, MD, Principal Investigator — Society Hill Reproductive Medicine
Locations (1):
- Society Hill Reproductive Medicine, Philadelphia, Pennsylvania, United States